CLINICAL TRIAL: NCT06561633
Title: The Influence Factors of Bispectral Index Values Increment Caused by Sugammadex Administration During Steady-state Anesthesia
Brief Title: The Influence Factors of Bispectral Index Values Increment Caused by Sugammadex
Status: Completed | Type: Observational
Sponsor: Jun Zhang (Other)
Responsible Party: Sponsor-Investigator, Jun Zhang, Professor, Fudan University
Organization: Fudan University (Other)
Other Study IDs: BIS-Sugammadex
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: BIS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Sugammadex administration — After surgery was completed while the train-of-four ratio was zero, a steady-state intravenous anesthesia was maintained to keep a BIS value within the range of 40-60 for at least 5 minutes. Patients received sugammadex 2 mg.kg-1 after completed surgery.
  Other Names: BIS monitor

SUMMARY:
Sugammadex administration may increase the bispectral index (BIS) values during general anesthesia. The purpose of this study was to investigate the influence factors leading to increase in BIS value caused by sugammadex administration when continuous use of general anesthetics.

DETAILED DESCRIPTION:
Sugammadex administration may increase the bispectral index (BIS) values during general anesthesia. The purpose of this study was to investigate the influence factors leading to increase in BIS value caused by sugammadex administration when continuous use of general anesthetics. Patients undergoing elective surgery were included in this study. After surgery was completed while the train-of-four ratio was zero, a steady-state intravenous anesthesia was maintained to keep a BIS value within the range of 40-60 for at least 5 minutes. Patients received sugammadex 2 mg.kg-1 after completed surgery. BIS values were recorded every minute and clinical signs of awaking was also noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients with American Society of Anesthesiologists (ASA) physical status Ⅰ - Ⅱ scheduled for elective surgery who agreed to participate and who signed the informed consent were included. Other inclusion criteria were age between 18 and 80 years and scheduled for elective non-cardiothoracic and non-neurological cancer surgery under general anesthesia (GA)

Exclusion Criteria:

* Known hypersensitivity to sugammadex; severe renal insufficiency (creatinine clearance < 30 ml.min-1); treatment with toremifene, flucloxacillin or fusidic acid in the pre-operative or immediate postoperative period; and neuropsychiatric disorders or treatment with a psychotropic agent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational cohort study was approved by the Institutional Review Board of the Fudan University Shanghai Cancer Center (No.2407-Exp042). Patients with ASA Ⅰ - Ⅱ scheduled for elective surgery who agreed to participate and who signed the informed consent were included.
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2024-08-20 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-14 (Actual)

PRIMARY OUTCOMES:
BIS value | 5 minutes
  BIS value at 5th min after sugammadex administration

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, Professor, Study Chair — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No